CLINICAL TRIAL: NCT00662129
Title: Phase II Trial of Albumin-Bound Paclitaxel in Combination With Gemcitabine and Bevacizumab in Patients With Metastatic Breast Cancer
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation, Gemcitabine, and Bevacizumab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0735; NCI-2009-00666 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000593581 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel + gemcitabine + bevacizumab (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline and after every other course, and then after completion of treatment.
  After completion of study treatment, patients are followed periodically for 5 years.
  Interventions: Biological: bevacizumab; Drug: gemcitabine hydrochloride; Drug: paclitaxel albumin-stabilized nanoparticle formulation

INTERVENTIONS:
Biological: bevacizumab
Drug: gemcitabine hydrochloride
Drug: paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine together with bevacizumab works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 6-month progression-free survival rate of patients with metastatic breast cancer treated with paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and bevacizumab.

Secondary

* To determine the overall survival of patients treated with this regimen.
* To determine the progression-free survival of patients treated with this regimen.
* To determine the confirmed response rate in patients treated with this regimen.
* To determine the duration of response in patients treated with this regimen.
* To determine the time to treatment failure in patients treated with this regimen.
* To determine the quality of life of patients treated with this regimen.

OUTLINE: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and after every other course, and then after completion of treatment.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed infiltrating breast cancer

  * Clinical evidence of metastatic disease
* Measurable disease, defined as at least one measurable lesion per RECIST criteria

  * No non-measurable disease only, defined as all other lesions, including small lesions (longest diameter < 2 cm) and truly non-measurable lesions, including any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Patients with HER-2/neu positive tumors, must have received prior treatment with trastuzumab (Herceptin®) or have a contraindication for trastuzumab
* No evidence of active brain metastasis, including leptomeningeal involvement, on MRI or CT scan

  * CNS metastasis controlled by prior surgery and/or radiotherapy allowed

    * Must be asymptomatic for ≥ 2 months with no evidence of progression prior to study entry
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Life expectancy ≥ 12 weeks
* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Total bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 mg/dL
* Urine protein:creatinine ratio < 1 or urinalysis < 1+ protein

  * Patients discovered to have ≥ 1+ proteinuria at baseline must demonstrate 24-hour urine protein < 1 g
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study therapy
* Able to complete questionnaires alone or with assistance
* No peripheral neuropathy > grade 1
* No history of allergy or hypersensitivity to albumin-bound paclitaxel, paclitaxel, gemcitabine hydrochloride, bevacizumab, albumin, drug product excipients, or chemically similar agents
* No stage III or IV invasive, non-breast malignancy within the past 5 years
* No other active malignancy, except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Patient must not be receiving other specific treatment for a prior malignancy
* No uncontrolled hypertension (i.e., blood pressure [BP] > 160/90 mm Hg on ≥ 2 occasions at least 5 minutes apart)

  * Patients who have recently started or adjusted antihypertensive medications are eligible providing that BP is < 140/90 mm Hg on any new regimen for ≥ 3 different observations in ≥ 14 days
* No bleeding diathesis or uncontrolled coagulopathy
* No hemoptysis within the past 6 months
* No prior arterial or venous thrombosis within the past 12 months
* No history of cerebrovascular accident
* No history of hypertensive crisis or hypertensive encephalopathy
* No abdominal fistula or gastrointestinal perforation within the past 6 months
* No serious non-healing wound, ulcer, or fracture
* No clinically significant cardiac disease, defined as any of the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Unstable angina
  * Cardiac arrhythmias not well controlled with medication
  * Myocardial infarction within the past 12 months
* No comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for study entry or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for metastatic disease

  * May have received one prior adjuvant chemotherapy regimen
* Prior neoadjuvant chemotherapy allowed

  * More than 6 months since prior adjuvant or neoadjuvant taxane (i.e., docetaxel or paclitaxel) therapy
* Prior hormonal therapy in either adjuvant or metastatic setting allowed
* More than 4 weeks since prior radiotherapy (except if to a non-target lesion only, or single dose radiation for palliation)

  * Prior radiotherapy to a target lesion is allowed provided there has been clear progression of the lesion since radiotherapy was completed
* More than 4 weeks since prior cytotoxic chemotherapeutic agent or investigational drug
* More than 2 weeks since prior and no concurrent acetylsalicylic acid, anticoagulants, or thrombolytic agents (except for once-daily 81 mg acetylsalicylic acid)
* More than 6 weeks since prior major surgery, chemotherapy, or immunologic therapy
* More than 1 week since prior minor surgery (e.g., core biopsy)

  * Placement of a vascular access device within 7 days is allowed
* More than 3 months since prior neurosurgery
* No concurrent treatment in a different clinical study in which investigational procedures are performed or investigational therapies are administered

  * Trials related to symptom management (Cancer Control) which do not employ hormonal treatments or treatments that may block the path of the targeted agents used in this study may be allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W. Northfelt, MD, FACP, Study Chair — Mayo Clinic
Locations (92):
- United States (92):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Northfelt DW, Dueck AC, Flynn TP, et al.: Phase II trial combining nab-paclitaxel (NP), gemcitabine (G), and bevacizumab (B) in patients (pts) with metastatic breast cancer (MBC): NCCTG N0735. [Abstract] J Clin Oncol 29 (Suppl 15): A-1126, 2011.

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel + Gemcitabine + Bevacizumab: Patients receive 125 mg/m^2 paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and 1000 mg/m^2 gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and 15 mg/kg bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Started | 50
Completed | 47
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Cancel prior to beginning treatment | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: One patient had a major violation (sequence of drugs was incorrect on Day 8 of Cycle 1), one patient canceled treatment prior to beginning treatment, and one patient was ineligible. The ineligible patient was included in the final analysis, whereas the two patients were excluded.
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 55.5 [27.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: The primary endpoint of this trial is the 6-month progression-free survival rate. A patient is considered to be a 6-month progression-free survivor if the patient is 6 months from registration without a documentation of disease progression (note, the patient need not be on study treatment at 6 months to be considered a success). The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated using the properties of the binomial distribution. Progression is defined using the RECIST Criteria, as at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: at 6 months
Population: The ineligible patient was included in the final analysis with participants who completed the study as specified in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: proportion of patients progression-free
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 48
proportion of patients progression-free | 0.792 [0.647 to 0.882]

2. Secondary Outcome: Overall Survival Time
Description: Overall Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier (1958).
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 48
months | 24.4 [18.2 to 29.3]

3. Secondary Outcome: PFS Time
Description: Progression-free survival time is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death. The distribution of time to progression will be estimated using the method of Kaplan-Meier (1958). Progression is defined using the RECIST Criteria, as at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 48
months | 11.2 [8.7 to 13.8]

4. Secondary Outcome: Confirmed Response (Complete or Partial Response) Rate
Description: A confirmed response is defined to be either a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations at least 8 weeks apart. The confirmed response rate (percentage) will be estimated by the number of confirmed responses in evaluable patients divided by the total number of evaluable patients multiplied by 100. The appropriate confidence interval will be calculated based on the binomial distribution.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients with CR or PR
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 48
percentage of patients with CR or PR | 70.8 [55.9 to 83.1]

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented. If a patient dies subsequent to the confirmed response without a documentation of disease progression, the patient will be considered to have had disease progression at the time of their death. In the case of a patient failing to return for evaluations before a documentation of disease progression, the patient will be censored for progression on the date of last evaluation. The distribution of duration of response will be estimated using the method of Kaplan-Meier (1958).
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 34
months | 9.7 [5.9 to 14.7]

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. If the patient is considered to be a major treatment violation or is taken off study as a non-protocol failure, the patient will be censored on the date they were removed from treatment. The distribution of time to treatment failure will be estimated using the method of Kaplan-Meier (1958). Progression is defined using the RECIST Criteria, as at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 48
months | 6.9 [5.2 to 8.5]

7. Secondary Outcome: Quality of Life, as Measure by the Mean Change in FACT-B TOI Score at Cycle 8
Description: Quality of life (QOL) as measured by the mean change (from baseline) in FACT-B (TOI) Trial Outcome Index at Cycle 8 (24 weeks). FACT-B was scored according to the published scoring (*) criteria with higher scores representing better QOL. The FACT-B TOI was the sum of the following FACT-B subscale/scale scores: physical (score range 0-28), functional (score range 0-28), and Breast Cancer Subscale (score range 0-40); range of the FACT-B TOI is 0-96 (the change scores have a possible range of -96 to 96). The mean change and 95% confidence interval are reported below. A one-sample t-test is used to compare the change from baseline to a value of 0.
  (*)= Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast (FACT-B) quality of life instrument. J Clin Oncol 1997;15:974-986.
Time Frame: From baseline to end of Cycle 8; Up to 24 weeks
Population: Of the participants evaluable for primary analysis, the Overall Number of Participants Analyzed reflects the number of subjects evaluable for this secondary outcome (with a FACT-B Trial Outcome Index score at baseline and at Cycle 8).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 27
units on a scale | -7.4 [-12.1 to -2.8]
Statistical Analysis 1: Comparison: Paclitaxel + Gemcitabine + Bevacizumab; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events are assessed 15 days prior to registration, and during the Active Monitoring Phase at each evaluation 3 days prior to each cycle of treatment and at the end of treatment; up to 2 years.
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 for adverse event monitoring and reporting. All graded adverse events are reported. Any participant whose adverse event(s) were assessed during the time frame specified above were included in the Adverse Events data tables below (i.e. All study participants excluding those who cancelled prior to beginning treatment as specified in the Participant Flow section).
Arm/Group | Paclitaxel + Gemcitabine + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 20/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Gemcitabine + Bevacizumab (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Amylase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Bilirubin increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 4 (6)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 10 (13)
Platelet count decreased (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Gemcitabine + Bevacizumab (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 42 (308)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Atrial flutter (Cardiac disorders) | 2 (5)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 11 (21)
Diarrhea (Gastrointestinal disorders) | 27 (88)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (8)
Mucositis oral (Gastrointestinal disorders) | 32 (95)
Nausea (Gastrointestinal disorders) | 37 (169)
Oral pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 24 (61)
Chest pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 5 (9)
Fatigue (General disorders) | 48 (449)
Fever (General disorders) | 23 (41)
Injection site reaction (General disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 4 (4)
Bladder infection (Infections and infestations) | 3 (5)
Catheter related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (6)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (3)
Alanine aminotransferase increased (Investigations) | 6 (9)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Bilirubin increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 12 (23)
Lymphocyte count decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 40 (153)
Platelet count decreased (Investigations) | 32 (105)
Weight loss (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 7 (11)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 34 (190)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (134)
Dizziness (Nervous system disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 37 (345)
Syncope (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 2 (3)
Protein urine positive (Renal and urinary disorders) | 20 (69)
Renal failure (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (152)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 30 (169)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 48 (454)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 12 (44)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 9 (11)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 6 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes